CLINICAL TRIAL: NCT06414512
Title: Optimizing the Dose of Flucytosine for the Treatment of Cryptococcal Meningitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Minnesota (Other)
Collaborators: Infectious Diseases Institute, Makerere University (Unknown); Mbarara University of Science and Technology (Other); Meningitis Foundation (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00017800; R01NS0863121 (Other: National Institutes of Health)
Record Dates: First submitted 2024-05-07; First posted 2024-05-16 (Actual); Results first posted 2025-08-27 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: Cryptococcal Meningitis
MeSH Terms: conditions — Meningitis, Cryptococcal | interventions — Flucytosine

STUDY DESIGN:
Intervention Model Description: Prospective, open-label trial to compare the efficacy and safety of lower doses of 5FC during induction therapy to historical controls with standard 5FC dosing. Historical controls drawn from the AMBITION trial will be used as a comparison group, selected weighted by inclusion/exclusion criteria, baseline characteristics and therapies received.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- control (Active Comparator): Historical controls drawn from the AMBITION trial will be used as a comparison group, selected weighted by inclusion/exclusion criteria, baseline characteristics and therapies received.
  Interventions: Drug: AMBITION trial control
- Low Dose Flucytosine (Experimental): HIV-infected persons in Uganda with cryptococcal meningitis
  Interventions: Drug: Flucytosine

INTERVENTIONS:
Drug: AMBITION trial control — Induction therapy for control group participants followed the 2018 WHO cryptococcal guidelines with 7 days of 5-FC 100mg/kg/day and 7 days of IV Amphotericin deoxycholate followed by 1200mg fluconazole/day for 7 days.
  Arms: control
Drug: Flucytosine — Participants in the trial will receive 60mg/kg/day of 5-FC in 3 divided doses for 10 days. Single-dose liposomal amphotericin (10mg/kg) is preferred, if available. Amphotericin B 0.7-1.0 mg/kg/day may be used if needed.
  Arms: Low Dose Flucytosine

SUMMARY:
Cryptococcal meningitis (CM) is a fungal infection that causes a severe syndrome of meningitis that is 100% fatal without antifungal therapy. Even with antifungal therapy, mortality rates remain high, especially in Africa where the ongoing HIV/AIDS pandemic leads to higher prevalence of cryptococcosis. Combination of amphotericin and flucytosine (5-FC) is the mainstay of therapy for the initial management of CM. Indeed, it has even been shown that effective delivery of these therapies in Africa can lower mortality rates by 90%.

This is a prospective open-label trial to compare the efficacy and safety of lower doses of 5FC during induction therapy to historical controls with standard 5FC dosing. Participants in the trial will receive 60mg/kg/day of 5-FC in 3 divided doses for 10 days. Single-dose liposomal amphotericin (10mg/kg) is preferred, if available. Amphotericin B 0.7-1.0 mg/kg/day may be used if needed. Historical controls drawn from the AMBITION trial will be used as a comparison group, selected weighted by inclusion/exclusion criteria, baseline characteristics and therapies received. Induction therapy for control group participants followed the 2018 WHO cryptococcal guidelines with 7 days of 5-FC 100mg/kg/day and 7 days of IV Amphotericin deoxycholate followed by 1200mg fluconazole/day for 7 days. The intervention group received single- dose liposomal amphotericin plus 5-FC and fluconazole 1200 mg/day.

All participants will receive fluconazole 1200mg/day during consolidation therapy from day 1 to 14 then 800mg/day from day 15 to 10 weeks, and 200mg/day after 10 weeks. All participants will receive lumbar punctures at diagnosis, day 3, day 5-7, day 10-14, and additionally as required for control of intracranial pressure and documentation of CSF sterilization. Controls from Ambition will be matched for the same LP windows. Therapeutic LPs conducted during the first week have a ~70% relative survival benefit.

ELIGIBILITY:
Inclusion Criteria:

* CSF cryptococcal antigen (CrAg) positive meningitis
* Ability and willingness to provide informed consent
* Willing to receive protocol-specified lumbar punctures

Exclusion Criteria:

* Age <18 years
* Inability to take enteral (oral or nasogastric) medicine
* Cannot or unlikely to attend regular clinic visits
* Receiving chemotherapy or corticosteroids
* Suspected Paradoxical immune reconstitution inflammatory syndrome (IRIS)
* Pregnancy or breastfeeding
* CrCl < 20 mL/minute
* Absolute neutrophil count <500 x10 6 cells/L
* Thrombocytopenia < 50,000 x 10 6 cells/L
* Patients with prior 5-flucytosine exposure >3 days in the 12 months prior to enrollment
* Any condition for which participation would not be in the best interest of the participant or that could limit protocol specified assessments.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2024-04-09 (Actual); Primary Completion 2024-10-02 (Actual); Study Completion 2024-10-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David B Meya, Principal Investigator — University of Minnesota; David R Boulware, Principal Investigator — University of Minnesota
Locations (2):
- Uganda (2):
  - Infectious Disease Institute, Mulago Hospital Complex, Kampala
  - Mbarara University of Science and Technology, Mbarara

REFERENCES:
- [Derived] Rutakingirwa MK, Skipper CP, Dai B, Wele A, Namombwe S, Mugabi T, Ndyetukira JF, Sadiq A, Kabahubya M, Chemusto L, Ahimbisibwe C, Nabbale S, Kandole TK, Muyise RCB, Kagimu E, Luggya T, Mulungi J, Jjunju S, Nicol MR, Stott KE, Kwizera R, Meya DB, Boulware DR, McHale TC; FLOOR trial team. Evaluating the Use of Lower Dose Flucytosine for the Treatment of Cryptococcal Meningitis: A Clinical Trial. Clin Infect Dis. 2025 Aug 7:ciaf432. doi: 10.1093/cid/ciaf432. Online ahead of print. PMID 40795226

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Controls were data drawn from another trial, not enrolled in this trial directly.
Period: Overall Study
Arm/Group | Control | Low Dose Flucytosine
Started | 171 | 48
Completed | 171 | 47
Not Completed | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | Low Dose Flucytosine | Total
Number analyzed (Participants) | 171 | 48 | 219
Age, Continuous [Mean (Inter-Quartile Range); unit: years] | 36 [30 to 42] | 40 [31 to 46] | 37 [32 to 44]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 70 | 26 | 96
  Male | 101 | 22 | 123
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Early Fungicidal Activity
Description: Rate of clearance of Cryptococcus from CSF.
Time Frame: 2 weeks
Population: The number analyzed are lower because not all enrolled had data for these outcomes.
Measure: Mean (Standard Deviation); unit: log10 CFU/mL/day
Arm/Group | Control | Low Dose Flucytosine
Number analyzed (Participants) | 97 | 44
log10 CFU/mL/day | 0.39 (0.27) | 0.28 (0.28)

2. Secondary Outcome: CSF Culture Sterility
Description: Cryptococcus is cleared or not from the cerebrospinal fluid
Time Frame: 18 weeks
Population: The number analyzed are lower because not all enrolled had data for these outcomes.
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Low Dose Flucytosine
Number analyzed (Participants) | 97 | 44
Participants | 60 | 25

3. Secondary Outcome: Mortality
Description: The proportion of participants who died after 16 weeks follow up
Time Frame: 16 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Low Dose Flucytosine
Number analyzed (Participants) | 171 | 48
Participants | 50 | 11

ADVERSE EVENTS:
Time Frame: 16 weeks
Arm/Group | Control | Low Dose Flucytosine
All-Cause Mortality (participants affected / at risk) | 50/171 | 11/48
Serious Adverse Events (participants affected / at risk) | 132/171 | 31/48
Other Adverse Events (participants affected / at risk) | 87/171 | 25/48
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control (N=171) | Low Dose Flucytosine (N=48)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
Acute Kidney Injury (Renal and urinary disorders) | 2 (2) | 4 (4)
Anemia (Blood and lymphatic system disorders) | 5 (5) | 2 (2)
Metabolic Encephalopathy (Metabolism and nutrition disorders) | 0 (0) | 3 (3)
Paradoxical CM IRIS (Infections and infestations) | 4 (4) | 4 (4)
Generalized tonic-clonic seizures (Nervous system disorders) | 0 (0) | 2 (2)
Other (General disorders) | 0 (0) | 3 (3)
CM Relapse (Infections and infestations) | 2 (2) | 6 (6)
URI Bronchitis/ Sinusitis (Infections and infestations) | 0 (0) | 1 (1)
Likely CM Persistence (Infections and infestations) | 0 (0) | 1 (1)
CNS Mass (Nervous system disorders) | 0 (0) | 2 (2)
Drug Induced Liver Injury (Hepatobiliary disorders) | 1 (1) | 0 (0)
Elevated Liver Enzymes (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hypoglycemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 7 (7) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 7 (7) | 0 (0)
Abnormal Increase in CSF QCC (Nervous system disorders) | 2 (2) | 0 (0)
Acute Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Acute Hypersensitivity Reaction (Immune system disorders) | 1 (1) | 0 (0)
Bacteremia/ Sepsis (Infections and infestations) | 2 (2) | 0 (0)
Clinical Deterioration (General disorders) | 3 (3) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 2 (2) | 0 (0)
Headache with Vomiting and Blurring (General disorders) | 1 (1) | 0 (0)
Intestinal Obstruction (Gastrointestinal disorders) | 2 (2) | 0 (0)
Neurologic Deterioration (Nervous system disorders) | 1 (1) | 0 (0)
Phlebitis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 0 (0)
Prolonged Hospitalization (Surgical and medical procedures) | 15 (15) | 0 (0)
Readmission (Surgical and medical procedures) | 25 (25) | 0 (0)
Recurrence of Symptoms (Infections and infestations) | 3 (3) | 0 (0)
Respiratory Distress (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 0 (0)
Severe scalp herpes zoster (Infections and infestations) | 1 (1) | 0 (0)
Tuberculosis (Infections and infestations) | 1 (1) | 0 (0)
Thrombophlebitis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Death, unknown cause (Investigations) | 29 (29) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control (N=171) | Low Dose Flucytosine (N=48)
Creatinine Grade 3 or Worse (Renal and urinary disorders) | 3 (3) | 1 (1)
Hemoglobin Grade 3 or Worse (Blood and lymphatic system disorders) | 17 (17) | 7 (7)
Elevated Liver Enzymes, Grade 3 or Worse (Hepatobiliary disorders) | 5 (5) | 3 (3)
Potassium Grade 3 or worse (Metabolism and nutrition disorders) | 7 (7) | 1 (1)
Hyponatremia Grade 3 or worse (Metabolism and nutrition disorders) | 7 (7) | 1 (1)
Leukopenia Grade 3 or worse (Blood and lymphatic system disorders) | 16 (16) | 5 (5)
Neutropenia Grade 3 or worse (Blood and lymphatic system disorders) | 23 (23) | 7 (7)
Thrombocytopenia (Blood and lymphatic system disorders) | 9 (9) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-03-22): https://cdn.clinicaltrials.gov/large-docs/12/NCT06414512/Prot_SAP_000.pdf
  • Informed Consent Form (2024-02-02): https://cdn.clinicaltrials.gov/large-docs/12/NCT06414512/ICF_001.pdf